CLINICAL TRIAL: NCT00992563
Title: A Dose-Escalation Study of AL-39324 Suspension Versus Lucentis® for the Treatment of Exudative Age-Related Macular Degeneration
Brief Title: WALTZ - Wet Age-Related Macular Degeneration (AMD) AL-39324 Treatment Examination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-023
Record Dates: First submitted 2009-10-07; First posted 2009-10-09 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Age Related Macular Degeneration
Keywords: wet age-related macular degeneration, exudative
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- AL-39324 Concentration Level A (Experimental): AL-39324 ophthalmic suspension, single intravitreal injection
  Interventions: Drug: AL-39324 ophthalmic suspension
- AL-39324 Concentration Level B (Experimental): AL-39324 ophthalmic suspension, single intravitreal injection
  Interventions: Drug: AL-39324 ophthalmic suspension
- AL-39324 Concentration Level C (Experimental): AL-39324 ophthalmic suspension, single intravitreal injection
  Interventions: Drug: AL-39324 ophthalmic suspension
- AL-39324 Concentration Level D (Experimental): AL-39324 ophthalmic suspension, single intravitreal injection
  Interventions: Drug: AL-39324 ophthalmic suspension
- AL-39324 Concentration Level E (Experimental): AL-39324 ophthalmic suspension, single intravitreal injection
  Interventions: Drug: AL-39324 ophthalmic suspension
- Lucentis (Active Comparator): Ranibizumab 10 mg/mL solution, single intravitreal injection
  Interventions: Drug: Ranibizumab 10 mg/mL

INTERVENTIONS:
Drug: AL-39324 ophthalmic suspension
  Arms: AL-39324 Concentration Level A; AL-39324 Concentration Level B; AL-39324 Concentration Level C; AL-39324 Concentration Level D; AL-39324 Concentration Level E
Drug: Ranibizumab 10 mg/mL
  Other Names: Lucentis®
  Arms: Lucentis

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and effects of investigational drug AL-39324 for the treatment of wet AMD.

DETAILED DESCRIPTION:
Following a single administration, patients will be followed for 6 months postinjection.

ELIGIBILITY:
Inclusion Criteria:

* Willing to give written informed consent, make the required study visits and follow instructions;
* The study eye:

  * must have a primary diagnosis of choroidal neovascularization (CNV) secondary to AMD;
  * lesion must be no larger than 30 mm2;
  * must have edema measuring greater than 340 μm;
  * must have a visual score between 73 and 34 letters, inclusive;
  * must be able to have clear picture taken of the back of the eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* The study eye must not have been treated for exudative AMD previously;
* The study eye must not have any other ocular disease, condition, infection, or recent surgery that would interfere with vision or examination of the back of the eye;
* The study eye must not have uncontrolled glaucoma;
* The study eye must not be missing a lens;
* Must not be taking any medication that is toxic to the lens;
* Must not be taking oral or ocular corticosteroids;
* Must not have an unstable or progressive condition that would interfere with study visits;
* Must not have allergies to any component of the test article or sensitivity to fluorescein dye;
* If female, must not be pregnant or nursing and must agree to adequate birth control;
* Must not be participating in another drug or device study within 30 days of screening for this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Incidence of targeted adverse events occurring in the study eye | Up to Day 7 after injection

SECONDARY OUTCOMES:
Mean change from baseline in central foveal thickness (CFT) at Month 1 | Baseline (Day 0), Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M. Kissner, Ph.D., Study Director — Alcon Research